CLINICAL TRIAL: NCT03087825
Title: Effect of Preoxygenation With Spontaneous Breathing or Noninvasive Positive Pressure Ventilation With or Without a Calibrated Leak. An Experimental Study in Healthy Volunteers
Brief Title: Preoxygenation Method With a Calibrated Leak
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: A15-D28-VOL.25
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-02

CONDITIONS: Preoxygenation; Non Invasive Ventilation

STUDY DESIGN:
Intervention Model Description: 2 groups : spontaneous breathing and non invasive pressure support ventilation 2 conditions : without inward air leak and with inward air leak
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- spontaneous breathing (Sham Comparator): preoxygenation through spontaneous breathing of 100% oxygen gas flow with or without an inward air leak
  Interventions: Procedure: preoxygenation without inward leak; Procedure: preoxygenation with inward leak
- pressure support ventilation (Active Comparator): preoxygenation through non invasive pressure support ventilation of 100% oxygen gas flow (inspiratory trigger sensitivity set at -2 l.min-1, the positive inspiratory support set at +6 cmH2O, the PEEP set at +5 cmH2O and the maximal airway pressure was limited at 15 cmH2O.) with or without an inward air leak
  Interventions: Procedure: preoxygenation without inward leak; Procedure: preoxygenation with inward leak

INTERVENTIONS:
Procedure: preoxygenation without inward leak — breathing a 100% inspired oxygen gas flow during 3 to 10 minutes
Procedure: preoxygenation with inward leak — breathing a 100% inspired oxygen gas flow during 3 to 10 minutes with an inward air leak made possible through a specific calibrated piece on the inspiratory branch

SUMMARY:
During preoxygenation, imperfect seal between the face mask and patient's face can induce an inward air leak decreasing its effectiveness. We assume that noninvasive ventilation could cancel the effect of the leak.

This is a prospective study. Healthy volunteers are randomised in cross-over between spontaneous breathing or noninvasive ventilation pressure support preoxygenation in the presence or absence of a calibrated leak on the inspiratory circuit.

DETAILED DESCRIPTION:
During preoxygenation, imperfect seal between the face mask and patient's face can induce an inward air leak decreasing its effectiveness. We assume that noninvasive ventilation could cancel the effect of the leak.

We planned an experimental study with healthy volunteers (residents in anesthesiology).

Healthy volunteers are randomised in cross-over between preoxygenation through spontaeous breathing or noninvasive ventilation pressure support preoxygenation in the presence or absence of a calibrated leak on the inspiratory circuit. The inspiratory fraction of oxygen is 100%. The exhaled gas (oxygen and carbon dioxide) are monitored.The subjects breathed through a mouthpiece (with a nose clip) connected to an anesthetic ventilator.

The primary endpoint is the time to achieve end expiratory fraction of oxygene of 90% or more.

The secondary endpoint is the proportion of subject with end expiratory fraction of oxygen of 90% or more after a 3 min period (recommended in clinical guidelines).

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* any pathological condition
* active tobaco

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
end expiratory fraction of oxygen | 10 minutes
  end expiratory fraction of oxygen measured in exhaled gas

CONTACTS AND LOCATIONS:
Overall Officials: jean-luc hanouz, m.D,ph.d, Principal Investigator — CHU de Caen and universite Caen Normandie
Locations (1):
- University Hospital of Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hanouz JL, Le Gall F, Gerard JL, Terzi N, Normand H. Non-invasive positive-pressure ventilation with positive end-expiratory pressure counteracts inward air leaks during preoxygenation: a randomised crossover controlled study in healthy volunteers. Br J Anaesth. 2018 Apr;120(4):868-873. doi: 10.1016/j.bja.2017.12.002. Epub 2018 Jan 17. PMID 29576128